CLINICAL TRIAL: NCT06292702
Title: Reduce Voiding Dysfunction After Laparoscopic Burch Colposuspension by Using Lateral Tension for the Anterior Vaginal Wall Before Cooper's Ligament Suspension in Stress Incontinence Women. (A Randomized Controlled Clinical Trial).
Brief Title: Reducing Early Urinary Disorders After Stress Incontinence Surgery: The Role of Vaginal Wall Tension.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Modified Burch Colposuspension
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence.; Burch colposuspension.; Voiding dysfunction.; Tension-free vaginal tape.; TVT, TOT, TVT-O.
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional laparoscopic Burch procedure (Experimental): Patients who were randomized to receive classic laparoscopic Burch colposuspension.
  Interventions: Procedure: Traditional Burch colposuspension
- Modified laparoscopic Burch procedure: (Experimental): Patients who were randomized to receive modified laparoscopic Burch colposuspension by applying lateral tension for the anterior vaginal wall before performing traditional anterior vaginal wall suspension toward Cooper's ligament.
  Interventions: Procedure: Modified Burch colposuspension

INTERVENTIONS:
Procedure: Traditional Burch colposuspension — Peforming two stitches between the anterior vaginal wall and Cooper's ligament.
  Arms: Traditional laparoscopic Burch procedure
Procedure: Modified Burch colposuspension — Performing lateral tension for the anterior vaginal wall towards the intersection point of the arcus tendineus and the lower edge of the pubic bone then performing two stitches between the anterior vaginal wall and Cooper's ligament.
  Arms: Modified laparoscopic Burch procedure:

SUMMARY:
The progress in surgical procedures for treating female stress urinary incontinence has led to the development of tension-free techniques such as the trans-obturator tape (TOT). Nonetheless, concerns regarding complications associated with the use of artificial mesh have sparked renewed interest in traditional retropubic suspension techniques (Burch). This study introduces a modified technique that creates lateral tension for the anterior vaginal wall before the conventional suspending to the Cooper ligament, limiting the tension on the urethra and reducing the risk of postoperative urinary voiding dysfunction with the same success rates. This technique offers the advantages of a tension-free procedure while still providing the benefits of retropubic suspension. Moreover, this modified technique eliminates the need for artificial mesh, reducing the risk of associated complications. This promising alternative offers effective support for the urethra and reduces postoperative emptying disorders. However, further research and studies are necessary to validate the long-term efficacy and safety of this modified technique.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial that aims to collect a sample within two years from the date of approval of the Scientific Research Council at Damascus University. The study will focus on a group of patients who will undergo a Burch colposuspension procedure, which is a surgical treatment for stress urinary incontinence. The patients will be randomly divided into two groups.

The first group will undergo a traditional Burch colposuspension, which involves lifting the vagina towards the Cooper ligament. The second group will receive a modified Burch colposuspension, which involves applying lateral tension for the anterior vaginal wall before the routine suspension on the Cooper ligament. The patients will then be followed for at least 3 months.

Data will be collected from the patients included in the study before the surgical operation, and then the patients will be followed up for at least three months after the surgery. The data will be compared between the two groups in terms of voiding dysfunction after surgery, which will be assessed according to International Consultation on Incontinence Questionnaire-Female Lower Urinary Tract Symptoms ICIQ_FLUTS and by assessing uroflowmetry, urinary retention, and post-void residual (PVR) urine.

Additionally, the recovery from stress incontinence will be compared by using The Patient's Global Impression of Improvement (PGI-I) and the stress test.

ELIGIBILITY:
Inclusion Criteria:

* The female patients with urinary incontinence are visiting the urology clinic due to a history of stress urinary incontinence, with failure of conservative treatment or non-compliance with treatment.

Exclusion Criteria:

* Patients refusing study participation.
* Contraindication to general anesthesia.
* Contraindication to laparoscopic surgery.
* Coexisting other type of urinary incontinence with urodynamic disturbance.
* Preoperative post-void residual urine.
* Previous pelvic irradiation.
* Concurrent anatomical deformity associated with genital prolapse, cystocele, or intrinsic sphincteric deficiency ( ISD ).

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Monosexual research (females with stress urinary incontinence)
Enrollment: 38 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Subjective voiding dysfunction after surgery, first evaluation | One week after surgery
  Voiding dysfunction will be assessed by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). It is composed of 12 questions, each question with a score from 0 to 4. Thus, the range of overall scores is from 0 to 16, 12, and 20 for filling, obstructive voiding, and incontinence scales, respectively. The total score range is from 0 to 48 for all types of voiding dysfunction after surgery
Urinary peak flow rate after surgery, first evaluation | One week after surgery
  Urinary peak flow rate will be determined by uroflowmetry, and divided into normal urinary flow rate for any value above or equal to 12 ml/sec, and abnormal urinary flow rate for any value under 12 ml/sec.
Residual urine after surgery, first evaluation | One week after surgery
  Residual urine will be assessed by ultrasound after voiding. All residual urine below 50 ml is considered insignificant and normal, while any residual urine above 50 ml is considered clinically significant and abnormal.
Urinary retention after surgery, first evaluation | One week after surgery
  Urinary retention will be assessed by clinical examination and ultrasound. It refers to the inability to void despite having a full bladder.
Subjective voiding dysfunction after surgery, second evaluation | One month after surgery
  Voiding dysfunction will be assessed by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). It is composed of 12 questions, each question with a score from 0 to 4. Thus, the range of overall scores is from 0 to 16, 12, and 20 for filling, obstructive voiding, and incontinence scales, respectively. The total score range is from 0 to 48 for all types of voiding dysfunction after surgery
Urinary peak flow rate after surgery, second evaluation | One month after surgery
  Urinary peak flow rate will be determined by uroflowmetry, and divided into normal urinary flow rate for any value above or equal to 12 ml/sec, and abnormal urinary flow rate for any value under 12 ml/sec.
Residual urine after surgery, second evaluation | One month after surgery
  Residual urine will be assessed by ultrasound after voiding. All residual urine below 50 ml is considered insignificant and normal, while any residual urine above 50 ml is considered clinically significant and abnormal.
Urinary retention after surgery, second evaluation | One month after surgery
  Urinary retention will be assessed by clinical examination and ultrasound. It refers to the inability to void despite having a full bladder.
Subjective voiding dysfunction after surgery, third evaluation | Three months after surgery
  Voiding dysfunction will be assessed by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF). It is composed of 12 questions, each question with a score from 0 to 4. Thus, the range of overall scores is from 0 to 16, 12, and 20 for filling, obstructive voiding, and incontinence scales, respectively. The total score range is from 0 to 48 for all types of voiding dysfunction after surgery
Urinary peak flow rate after surgery, third evaluation | Three months after surgery
  Urinary peak flow rate will be determined by uroflowmetry, and divided into normal urinary flow rate for any value above or equal to 12 ml/sec, and abnormal urinary flow rate for any value under 12 ml/sec.
Residual urine after surgery, third evaluation | Three months after surgery
  Residual urine will be assessed by ultrasound after voiding. All residual urine below 50 ml is considered insignificant and normal, while any residual urine above 50 ml is considered clinically significant and abnormal.
Urinary retention after surgery, third evaluation | Three months after surgery
  Urinary retention will be assessed by clinical examination and ultrasound. It refers to the inability to void despite having a full bladder.

SECONDARY OUTCOMES:
Subjective recovery from urinary incontinence, first evaluation | one week after surgery
  Subjective recovery from urinary incontinence will be assessed by the Patient's Global Impression of Improvement (PGI-I). It is an instrument designed to measure a patient's interpretation of symptom changes following intervention.
  The patient enters his answer on a 7-point scale scored as (1) "very much better," to (7) "very much worse."
Objective recovery from urinary incontinence, first evaluation | one week after surgery
  Objective recovery will be assessed by a urinary stress test by filling the bladder and telling the patient to make an effort and cough and repeat it three times.
  The negative test is considered an objective recovery
Subjective recovery from urinary incontinence, second evaluation | One month after surgery
  Subjective recovery from urinary incontinence will be assessed by the Patient's Global Impression of Improvement (PGI-I). It is an instrument designed to measure a patient's interpretation of symptom changes following intervention.
  The patient enters his answer on a 7-point scale scored as (1) "very much better," to (7) "very much worse."
Objective recovery from urinary incontinence, second evaluation | One month after surgery
  Objective recovery will be assessed by a urinary stress test by filling the bladder and telling the patient to make an effort and cough and repeat it three times.
  The negative test is considered an objective recovery
Subjective recovery from urinary incontinence, third evaluation | three months after surgery
  Subjective recovery from urinary incontinence will be assessed by the Patient's Global Impression of Improvement (PGI-I). It is an instrument designed to measure a patient's interpretation of symptom changes following intervention.
  The patient enters his answer on a 7-point scale scored as (1) "very much better," to (7) "very much worse."
Objective recovery from urinary incontinence, third evaluation | three months after surgery
  Objective recovery will be assessed by a urinary stress test by filling the bladder and telling the patient to make an effort and cough and repeat it three times.
  The negative test is considered an objective recovery

CONTACTS AND LOCATIONS:
Overall Officials: Samir M Enzawi, M.D, Ph.D, Study Director — dr.enzsamir58@gmail.com
Locations (1):
- Damascus university, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Natale F, La Penna C, Saltari M, Piccione E, Cervigni M. Voiding dysfunction after anti-incontinence surgery. Minerva Ginecol. 2009 Apr;61(2):167-72. PMID 19255563
- [Result] Steele SS, Bailly GG. Choosing the right sling for your patient. Can Urol Assoc J. 2017 Jun;11(6Suppl2):S132-S134. doi: 10.5489/cuaj.4635. PMID 28616112
- [Result] Sassani JC, Artsen AM, Moalli PA, Bradley MS. Temporal Trends of Urogynecologic Mesh Reports to the U.S. Food and Drug Administration. Obstet Gynecol. 2020 May;135(5):1084-1090. doi: 10.1097/AOG.0000000000003805. PMID 32282600
- [Result] Karlovsky ME. How to Avoid and Deal with Pelvic Mesh Litigation. Curr Urol Rep. 2016 Aug;17(8):55. doi: 10.1007/s11934-016-0613-3. PMID 27287606
- [Result] Barr SA, Thomas A, Potter S, Melick CF, Gavard JA, McLennan MT. Incidence of successful voiding and predictors of early voiding dysfunction after retropubic sling. Int Urogynecol J. 2016 Aug;27(8):1209-14. doi: 10.1007/s00192-016-2972-1. Epub 2016 Feb 19. PMID 26894607
- [Result] Valdevenito JP, Mercado-Campero A, Naser M, Castro D, Ledesma M, Arribillaga L. Voiding dynamics in women with urinary incontinence but without voiding symptoms. Neurourol Urodyn. 2020 Nov;39(8):2223-2229. doi: 10.1002/nau.24475. Epub 2020 Aug 7. PMID 32767826